CLINICAL TRIAL: NCT02607904
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Pharmacokinetic Trial in 2 Parallel Groups to Investigate Possible Drug-drug Interactions Between Stiripentol or Valproate and GWP42003-P in Patients With Epilepsy
Brief Title: An Open-label Extension Trial to Investigate Possible Drug-drug Interactions Between Stiripentol or Valproate and Cannabidiol in Patients With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWEP1447 Open-label Extension; 2015-002939-18 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Epilepsy
Keywords: Cannabidiol; GWP42003-P; Epidiolex; Stiripentol; Valproate
MeSH Terms: conditions — Epilepsy | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GWP42003-P (Experimental): Administered orally, twice daily (morning and evening), commencing with titration of 100 mg/mL GWP42003-P to 20 mg/kg/day over 10 days in a blinded manner (i.e., only participants taking placebo in the blinded phase will up-titrate; doses will remain unchanged for those taking GWP42003-P in the blinded phase).
  Participants remain on the maintenance dose for the remainder of the 48-week treatment period, until early withdrawal or at an early study conclusion date defined by the sponsor. However, investigators may subsequently decrease or increase the participant's dose (to a maximum of 30 mg/kg/day) until the optimum dose is found.
  Dosing is tapered (10% each day) for participants who do not immediately continue to use GWP42003-P once market authorization is granted, or for those who withdraw early.
  Interventions: Drug: GWP42003-P

INTERVENTIONS:
Drug: GWP42003-P — Clear, colorless to yellow solution containing cannabidiol (CBD) dissolved in the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring.
  Other Names: Cannabidiol; CBD; Epidiolex

SUMMARY:
This trial consists of 2 parts: a double-blinded phase and an open-label extension phase. The open-label extension phase only will be described in this record. All participants will receive the same dose of GWP42003-P. However, investigators may subsequently decrease or increase the participant's dose until the optimal dose is found.

ELIGIBILITY:
Note: Participants who enroll in France or Sweden must be aged 18-55 years.

Key Inclusion Criteria:

* Participant must have a documented magnetic resonance imaging/computerized tomography of the brain that ruled out a progressive neurologic condition.

Key Exclusion Criteria:

* Participant has clinically significant unstable medical conditions other than epilepsy.
* Participant has a history of symptoms related to a drop in blood pressure due to postural changes (e.g., dizziness, light-headedness, blurred vision, palpitations, weakness, syncope).
* Participant has any history of suicidal behavior or any suicidal ideation of type 4 or 5 on the C-SSRS in the last month.
* Participant is currently using felbamate and has been taking it for less than 12 months prior to screening visit of the blinded phase of the trial.
* Participant is currently using or has in the past used recreational or medicinal cannabis, or synthetic cannabinoid-based medications (including Sativex®) within the 3 months prior to trial entry.
* Participant has any known or suspected history of any drug abuse or addiction.
* Participant is unwilling to abstain from recreational or medicinal cannabis, or synthetic cannabinoid-based medications (including Sativex) for the duration for the trial.
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients of the Investigational Medicinal Product (IMP), e.g., sesame oil.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Number of participants who experienced an adverse event. | Up to 48 weeks.
  The number of participants who experienced an adverse event during the trial is presented.

SECONDARY OUTCOMES:
Number of participants with a clinically significant change in 12-lead electrocardiogram (ECG). | Up to 48 weeks.
  The number of participants with a clinically significant change in ECG is presented.
Number of participants with a clinically significant change in serum biochemistry. | Up to 48 weeks.
  The number of participants with a clinically significant change in serum biochemistry is presented.
Number of participants with a clinically significant change in hematology. | Up to 48 weeks.
  The number of participants with a clinically significant change in hematology is presented.
Number of participants with a clinically significant change in urinalysis. | Up to 48 weeks.
  The number of participants with a clinically significant change in urinalysis is presented.
Number of participants with a clinically significant change in vital signs. | Up to 48 weeks.
  The number of participants with a clinically significant change in vital signs (systolic blood pressure, diastolic blood pressure, pulse rate) is presented.
Number of participants with a clinically significant change in physical examination. | Up to 48 weeks.
  The number of participants with a clinically significant change in physical examination is presented.
Number of participants with a treatment-emergent suicidality flag. | Up to 48 weeks.
  Suicidality was assessed using the Columbia-Suicide Severity Rating Scale (C-SSRS). The number of participants with a treatment-emergent flag is presented.
Seizure frequency by subtype. | Up to 48 weeks.
  The frequency of each subtype of seizure at baseline and end of treatment is presented.
Number of participants with a treatment-emergent finding indicative of drug abuse liability. | Up to 48 weeks.
  Abuse liability was assessed through monitoring of triggering adverse events of interest and study medication accountability discrepancies. Any findings were assigned to an appropriate classification by the investigator. The number of participants with a treatment-emergent finding indicative of drug abuse liability is presented.

CONTACTS AND LOCATIONS:
Locations (5):
- SEIN - Epilepsy Institute in the Netherlands Foundation, Zwolle, Netherlands
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No